CLINICAL TRIAL: NCT06242171
Title: Prognostic Indices of Atheromatosis Severity and Coronary Artery Bypass Surgery Outcomes for Patients With Coronary Artery Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Onassis Cardiac Surgery Centre (Other)
Responsible Party: Principal Investigator, Aikaterini Gavalaki, Research Fellow, Onassis Cardiac Surgery Centre
Other Study IDs: 697/20.10.2020
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Atheromatosis
Keywords: coronary sinus sampling; coronary artery bypass graft surgery
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary artery disease is a multifactorial disease. Traditional risk factors, such as obesity, diabetes, hypertension, stimulate the onset of an inflammatory process in the prone vessel and perivascular adipose tissue, which has not yet been clarified and is still being investigated.

Coronary artery bypass grafting is an effective treatment of coronary artery disease, which has been shown to prolong survival. Perioperative analysis of the myocardial metabolic profile helps to identify appropriate markers and metabolites associated with early myocardial damage. This, in turn, helps to improve risk stratification by better understanding the mechanisms of the disease processes, in order to prevent postoperative myocardial infarction and its associated complications. Such indicators, which are related to the diagnosis and severity of coronary artery disease, as well as the prognosis of coronary artery bypass grafting, have been separately studied before, in the peripheral blood of patients with coronary artery disease, in healthy vascular tissues, such as mammary artery, compared to atherosclerotic tissue from the coronary artery, as well as in the epicardial adipose tissue, intraoperatively.

The aim of the proposed study is to investigate and evaluate metabolic factors and biomarkers preoperatively, intraoperatively and postoperatively, in patients undergoing coronary artery bypass grafting and their prognostic value regarding a) the severity of coronary artery disease (Gensini score, ejection fraction, acute coronary syndrome) and b) the outcome of surgery (indications of myocardial damage and / or infarction, low cardiac output syndrome and use of intraortic balloon pump, atrial fibrillation, 30-day mortality).

DETAILED DESCRIPTION:
This is a prospective study, which will include 90 patients with diagnosed symptomatic coronary artery disease, who are scheduled to undergo coronary artery bypass surgery at the Onassis Cardiac Surgery Center. Patients with other cardiovascular diseases (valvular pathologies or aortic diseases) will not be included in the study.

A) Upon admission in hospital, patients will be informed and will sign their consent to participate in the research protocol. Subsequently, a complete medical history will be obtained, including risk factors, comorbidities, and medical treatment. Gensini score of coronary artery disease severity, ejection fraction, and history of acute coronary syndrome will also be recorded.

B) Preoperatively, a blood sample will be taken from a peripheral vein, part of which will be stored in RNA preservation tubes, and another part will be centrifuged in the Biochemistry Laboratory for plasma preservation.

C) Intraoperatively, and in chronological order:

Blood samples will be taken through the coronary sinus catheter just before initiating extracorporeal circulation, divided into four parts: 1) in RNA preservation tube, 2) in a tube for plasma isolation, 3) in a tube for direct biochemical analysis (TnI, NT-proBNP, LDH), and 4) in a blood gas analyzer for pO2, pCO2, SpO2, Lactate acid, Hgb calculation.

Tissue samples will be taken from the harvested internal mammary artery, atheroma of the coronary vessel, whenever possible and epicardial adipose tissue.

Blood sample through the coronary sinus catheter immediately after extracorporeal circulation, divided into two parts: 1) in a tube for direct biochemical analysis, and 2) in a blood gas analyzer for pO2, pCO2, SpO2, Lactate acid, Hgb calculation.

Simultaneously, at the same time points, blood samples will be taken from the radial or brachial artery before and after extracorporeal circulation, and analyzed for blood gases.

D) Postoperatively, a peripheral blood sample will be taken from the patient on the day of discharge; one part will be stored in RNA preservation tubes and another part centrifuged in the Biochemistry Laboratory for plasma preservation. In addition, intraoperative data (extracorporeal circulation duration, aortic cross-clamp time) and intervention outcome data (maximum troponin value and corresponding time, postoperative ejection fraction, atrial fibrillation event, intra-aortic pump placement, ICU stay duration, hospital stay duration, 30-day mortality) will be recorded.

E) All whole blood, plasma, and tissue samples will be immediately stored at -80°C, grouped for each case, until sent to the Laboratory of Biological Chemistry at the University of Athens for detection and quantification of indicators such as extracellular matrix metalloproteinases (MMP-2, MMP-9, TIMP1, TIMP2), cytokines (IFNγ, IL-2, IL-4, IL-5, IL-6), and microRNA expression.

F) After data collection, statistical analysis and correlation of various parameters measured in the coronary vessel, epicardial fat, patient's serum, and blood from the coronary sinus will be performed: 1) with the severity of coronary artery disease (Gensini score), and 2) with the short-term surgery outcome. Differences in the expression of study parameters between the coronary artery and internal mammary artery of the same patient will also be highlighted. These findings aim to identify new biomarkers of coronary artery disease and clarify the role of epicardial fat in the atheromatous process.

ELIGIBILITY:
Inclusion Criteria: Symptomatic coronary artery disease requiring surgical revascularisation

-

Exclusion Criteria:

Severe comorbidities; renal or liver failure, severe autoimmune disease Combined surgical procedures (valve surgery, aortic procedures, carotid surgery)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that are scheduled to have coronary artery bypass graft surgery in Onassis Cardiac Surgery Centre
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic and molecular indices identified in coronary sinus and peripheral blood, as well as in epicardial, coronary artery and internal mammary artery tissue | 3 years
  Correlation of the indices identified/ calculated with coronary artery disease severity and CABG outcome

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Perreas, MD, PhD, Study Director — Onassis Cardiac Surgery Centre
Locations (1):
- Onassis Cardiac Surgery Centre, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided